CLINICAL TRIAL: NCT00421044
Title: An Open-label, Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Patupilone in Patients With Advanced Solid Tumors and Varying Degrees of Hepatic Function
Brief Title: A Study of Patupilone in Patients With Advanced Solid Tumors and Varying Degrees of Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2121E1; NCT00478920 (obsolete NCT alias)
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Advanced Malignancies; Tumors
Keywords: EPO; Patupilone; Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — epothilone B

ARMS (3):
- Arm A (Normal liver function) (Experimental)
  Interventions: Drug: Patupilone/EPO906
- Arm B (Mild liver dysfunction) (Experimental)
  Interventions: Drug: Patupilone/EPO906
- Arm C (Moderate liver dysfunction) (Experimental)
  Interventions: Drug: Patupilone/EPO906

INTERVENTIONS:
Drug: Patupilone/EPO906

SUMMARY:
Patients who participated in the core EPO2121 study and did not clinically progress may participate in this extension protocol to further evaluate the safety, tolerability, and efficacy of patupilone.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the core study is required for participation in the extension.
* 18 years of age or older
* World Health Organization (WHO) Performance Status score of: 0 - you are fully active and more or less as you were before your illness; 1 - you cannot carry out heavy physical work, but can do anything else; or 2 - you are up and about more than half the day, you can look after yourself, but are not well enough to work.
* Life expectancy of 3 months or more
* Patients with measurable or evaluable disease who have histologically documented advanced solid tumor and who have progressed after systemic therapy or for whom standard systemic therapy does not exist

Exclusion Criteria:

* Severe and/or uncontrolled medical disease
* Known diagnosis of human immunodeficiency virus (HIV) infection
* Presence of any other active or suspected acute or chronic uncontrolled infection
* Severe cardiac insufficiency, with uncontrolled and/or unstable cardiac or coronary artery disease
* History of another malignancy within 5 years prior to study entry, except for curatively treated non-melanotic skin cancer or cervical cancer in situ

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2006-05; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability in patients with hepatic impairment will be assessed by adverse events (AEs), serious adverse events (SAEs) and out of range lab values | at completion of the study
To evaluate the preliminary anti-tumor activity which will be assessed by radiological scans every 6 weeks | at completion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (3):
- United States (3):
  - University of California San Diego/Moores Cancer Center, La Jolla, California
  - Institute for Drug Development Cancer Therapy & Research Center/The University of Texas Health Science Center, San Antonio, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas